CLINICAL TRIAL: NCT03091179
Title: The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Short Laryngologic Surgical Procedures.
Brief Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) and Short Laryngologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vladimir Nekhendzy, Clinical Professor of Anesthesiology and Otolaryngology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 39202
Record Dates: First submitted 2017-03-05; First posted 2017-03-27 (Actual); Results first posted 2019-07-17 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Laryngologic Surgical Procedures
Keywords: airway management; high flow nasal oxygen; high flow nasal cannula; THRIVE
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- THRIVE (Experimental): high flow nasal oxygen
  Interventions: Device: THRIVE
- Endotracheal tube (Active Comparator): tracheal intubation
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: THRIVE — active nasal oxygen delivery system
  Arms: THRIVE
Device: Endotracheal tube — a plastic tube for mechanical ventilation
  Arms: Endotracheal tube

SUMMARY:
The purpose of this study is to investigate whether selected, short laryngologic surgical procedures can be safely and potentially more effectively performed without the use of endotracheal tube or jet ventilation, under completely tubeless conditions. The patient's gas exchange will be supported by rapid insufflation of high-flow oxygen through specialized nasal cannulae: the so called Transnasal Humidified Rapid- Insufflation Ventilatory Exchange (THRIVE).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for short, non-laser laryngologic surgery

Exclusion Criteria:

1. Patients with significantly decreased myocardial function (ejection fraction < 50%)
2. Patients with abnormal cardiac rhythm and conduction abnormalities, except for patients with isolated, asymptomatic premature atrial and ventricular contractions.
3. Patients with significant peripheral vascular disease, such as those with the symptoms of intermittent claudication.
4. Patients with known significant cerebrovascular disease, such as history of cerebrovascular accidents (CVAs) and transient ischemic attacks (TIAs).
5. Patients with significant renal insufficiency, as manifested by estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2.
6. Patients with electrolyte (K+, Ca++) abnormalities, as determined by the lab values outside of a normal range.
7. Patients with the history or symptoms of increased intracranial pressure or reduced intracranial compliance (e.g. headaches, nausea and vomiting, visual changes, mental changes).
8. Patients with skull base defects.
9. Patients with pulmonary hypertension who have pulmonary artery pressures above the normal range.
10. Patients with significant chronic obstructive or restrictive lung diseases, as manifested by known history of baseline chronic hypoxia and/or hypercapnia, and/or baseline room air SpO2 < 95%.
11. Obese patients with BMI above 35 kg/m2.

13. Patients with severe and poorly controlled gastroesophageal reflux disease despite medical treatment.

14. Patients with hiatal hernia and full stomach patients. 15. Patient's refusal to participate in the study. 16. Patients who do not understand English or mentally handicapped. 17. Pregnant or breastfeeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Nekhendzy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nekhendzy V, Saxena A, Mittal B, Sun E, Sung K, Dewan K, Damrose EJ. The Safety and Efficacy of Transnasal Humidified Rapid-Insufflation Ventilatory Exchange for Laryngologic Surgery. Laryngoscope. 2020 Dec;130(12):E874-E881. doi: 10.1002/lary.28562. Epub 2020 Feb 20. PMID 32078170

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Endotracheal tube or Supraglottic jet ventilation
Period: Overall Study
Arm/Group | THRIVE | Control Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THRIVE | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.42) | 55.2 (17.29) | 53.1 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Average Oxygen Saturation by Pulse Oximetry (SpO2) (Primary Anesthesia Outcome)
Time Frame: intraoperative (up to one hour)
Measure: Mean (Standard Deviation); unit: percentage of saturation (SpO2)
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
percentage of saturation (SpO2) | 93 (5.66) | 98.7 (1.57)
Statistical Analysis 1: Comparison: THRIVE vs Control Group; Test type: Equivalence — P value was calculated using the means and standard deviations for each of the patient characteristics; p = 0.006, t-test, 2 sided

2. Primary Outcome: Time to Awakening From Anesthesia (Primary Anesthesia Outcome)
Description: time from end of surgery to responding to commands/extubation
Time Frame: intraoperative (up to 20 min)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
minutes | 10.3 (4.0) | 9.4 (3.4)

3. Primary Outcome: Suspension Time (Primary Surgical Outcome)
Description: Time required for the surgeon to position the patient's head and expose the surgical field for surgery using operating laryngoscope
Time Frame: intraoperative (up to 5 min)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
minutes | 1.8 (1.1) | 4.3 (2.1)

4. Primary Outcome: Number of Suspension Repositioning Maneuvers (Primary Surgical Outcome)
Description: Number of attempts required for the surgeon to reposition the patient's head for optimal surgical exposure using operating laryngoscope
Time Frame: intraoperative (up to 5 min)
Measure: Mean (Standard Deviation); unit: maneuvers
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
maneuvers | 0.4 (0.52) | 1.7 (0.95)

5. Primary Outcome: Duration of Surgery (Primary Surgical Outcome)
Time Frame: intraoperative (up to one hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
minutes | 19.1 (10.82) | 20.9 (8.85)

6. Secondary Outcome: Alertness
Description: Time required for the patient to become fully alert and oriented per standard recovery room evaluation
Time Frame: Recovery room admission (up to 30 min following admission to recovery room)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
minutes | 4.3 (6.3) | 4.8 (7.4)

7. Secondary Outcome: Recovery Room Time
Time Frame: Up to 2 hours after procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
minutes | 65.7 (43.41) | 77.7 (42.84)

8. Secondary Outcome: Numerical Pain Rating Scores
Description: A score from 0 to 10, higher scores corresponding to higher pain
Time Frame: Recovery room admission and discharge (up to 2 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
score on a scale
  recovery room admission | 1.3 (1.95) | 3.7 (2.91)
  recovery room discharge | 0.9 (1.29) | 2.7 (1.77)

9. Secondary Outcome: Opioid Consumption
Description: Total oral opioid consumption in morphine milligram equivalents
Time Frame: Recovery room admission and discharge (up to 2 hours)
Measure: Mean (Standard Deviation); unit: MME: morphine milligram equivalents
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
MME: morphine milligram equivalents | 8.8 (11.0) | 22.5 (22.1)

10. Secondary Outcome: Change in Voice Handicap Index (VHI)
Description: numerical scale, range from 0 to 40, with higher scores corresponding to worse outcome
Time Frame: Preoperative assessment and one month after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
score on a scale
  preoperative | 12.8 (12.63) | 22.7 (12.06)
  one month after surgery | 7.6 (12.19) | 13.6 (13.22)

11. Secondary Outcome: Quality of Recovery
Description: 15-question survey, with each question scored from 0 to 10. Overall range 0-150, higher scores correspond to better outcome.
Time Frame: One week after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Control Group
Number analyzed (Participants) | 10 | 10
score on a scale | 142.5 (15.7) | 131.2 (17.9)

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | THRIVE | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03091179/SAP_000.pdf
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03091179/Prot_001.pdf